CLINICAL TRIAL: NCT01620463
Title: A Randomised, Double-blind, Single-centre, Placebo-controlled, Ascending Single s.c. Dose, Sequential Group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC 90-1170 in Healthy Japanese Male Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Liraglutide in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1326
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 90-1170 (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Single dose administered subcutaneously at four different dose levels: 2.5, 5.0, 10.0 and 15.0 mcg/kg. Following completion of each dose group, an evaluation will be performed to allow progression to the next dose group
  Other Names: NNC 90-1170
  Arms: NNC 90-1170
Drug: placebo — Single dose administered subcutaneously at four different dose levels: 2.5, 5.0, 10.0 and 15.0 mcg/kg. Following completion of each dose group, an evaluation will be performed to allow progression to the next dose group
  Arms: Placebo

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to assess the safety and tolerability of NNC 90-1170 (liraglutide) in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 27 kg/m^2, inclusive

Exclusion Criteria:

* Clinically relevant abnormalities of physical examination, laboratory values, vital signs or ECG findings at the screening, as judged by the Investigator or Sub-Investigator
* Presence of acute or chronic illness sufficient to invalidate the subject's participation in the study or to make it unnecessarily hazardous, as judged by the Investigator
* Blood pressure in supine position at the screening, after resting for 5 min, outside the ranges 90-150 mmHg systolic or 40-90 mmHg diastolic
* Heart rate in supine position at the screening, after resting for 5 min, outside the range 40-100 beats/min
* Alcohol intake within 48 hours prior to the screening
* Hepatitis B surface antigen, Hepatitis C antibodies or HIV (human immunodeficiency virus) antibodies positive
* Clinically relevant abnormal history or physical findings at the screening, which could interfere with the objectives of the study or the safety of the subject's participation, as judged by the Investigator
* History of significant allergy or hypersensitivity
* Known or suspected allergy to trial product or related products
* History of drug or alcohol abuse
* Smoking 10 cigarettes or more, or the equivalent, per day and is unwilling to refrain from smoking during 3 days prior to dosing and during the confinement period

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2002-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Body weight
Vital signs (Blood pressure)
Vital signs (Pulse rate)
ECG (ElectroCardioGram)
Adverse events

SECONDARY OUTCOMES:
Area under the plasma NNC 90-1170 curve
Maximum plasma NNC 90-1170 concentration, Cmax
Time to maximum plasma NNC 90-1170 concentration, tmax
Terminal elimination half-life, t1/2
24-hour glucose profile in serum
24-hour insulin profile in serum
24-hour glucagon profile in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Result] Kageyama S, Hirao K, Shimizu A, Matsumura Y, Zdravkovic M, Rasmussen MF, Irie S. Tolerability, pharmacokinetics, and pharmacodynamics of liraglutide, long-acting human GLP-1 analogue - Phase 1 studies in Japanese healthy subjects with type 2 diabetes. Endocrinology and Diabetology 2007; 24 (6): 95-104
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com